CLINICAL TRIAL: NCT06546514
Title: The Effect of Breath Exercise Training Given to Patients Undergoing Surgery in the General Surgery Clinic on Postoperative Pain, Anxiety, and Nausea-Vomiting
Brief Title: The Impact of Breath Exercise Training on Postoperative Pain, Anxiety, and Nausea-Vomiting in General Surgery Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Gamze BULUT, Principal Investigator, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Gamze
Record Dates: First submitted 2024-08-07; First posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Postoperative Pain, Acute; Postoperative Nausea and Vomiting; Patient Relations, Nurse
Keywords: Postoperative Pain; Anxiety; Nausea-Vomiting; Nurse; Breathing Exercise; General Surgery
MeSH Terms: conditions — Pain, Postoperative; Postoperative Nausea and Vomiting; Anxiety Disorders | interventions — Breathing Exercises

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Grup 1 (Experimental): the group that performed breathing exercises
  Interventions: Other: Breath Exercise
- Grup 2 (No Intervention): the group that did not perform breathing exercises

INTERVENTIONS:
Other: Breath Exercise — It was provided by the researcher that the patients performed 5 repetitions of 10 breathing exercises every 3 hours a day, between 09:00am and 21:00pm, 1 day before the surgery, on the day of surgery and on the first day after surgery.
  Arms: Grup 1

SUMMARY:
This study was conducted to determine the effect of breath exercise on post-operative anxiety level, pain, and nausea-vomiting after general surgery. This was a randomized, controlled experimental study. The sample comprised 149 patients who underwent laparoscopic cholecystectomy and hernia (control:73; experimental:76). One day before the operation, the participants in the experimental group were given breathing exercise training, and they were applied 5 times a day for 10 repetitions until the 30th day after the operation.

DETAILED DESCRIPTION:
Today, surgical treatment is one of the areas where technological methods are frequently applied in the treatment of diseases and the recovery process of patients. Problems such as pain, nausea, vomiting, fear and anxiety occur after surgery, and these situations negatively affect the patient's comfort, quality of life, recovery and satisfaction; they also cause the length of hospital stay and the time allocated to nursing care to be extended and the cost to increase. Pain is a frequently seen symptom in the postoperative period. Approximately 86% of patients experience pain to varying degrees during this period. Prolonged postoperative pain paves the way for the development of various physiopathological responses such as immobility, increased oxygen consumption, atelectasis, deep vein thrombosis, tachycardia, hypertension, decreased stomach and intestinal motility, increased blood sugar, urinary retention and delayed wound healing. Anxiety plays an important role in the increase and decrease of pain after surgical intervention. Studies have determined that pain in the preoperative period increases the level of anxiety and that this situation lowers the pain threshold. Effectively managed and controlled postoperative pain; It reduces anxiety levels and facilitates keeping life parameters at an optimal level after surgical intervention.

Postoperative nausea and vomiting are seen in 20-30% of patients after general anesthesia and are the second most common complaint after pain, and this rate increases to 80% in high-risk groups. Despite antiemetic and analgesic drugs, postoperative nausea, vomiting and pain continue to be an important problem for patients today. Although postoperative nausea and vomiting is not a life-threatening complication, it is a condition that makes recovery from anesthesia difficult, causes fluid-electrolyte imbalance, increases the risk of aspiration, causes stress in patients, causes tension in the suture line and prolongs the discharge period. Many different pharmacological approaches have been developed to minimize postoperative nausea, vomiting and pain. However, the side effects of traditional antiemetics and analgesics and the high cost of drugs have increased the interest in the use of non-pharmacological methods.

Breathing exercises can be used as an effective, simple and cost-effective non-pharmacological approach to prevent or reduce the occurrence of postoperative complications. In addition, it has been shown in the literature that it also increases physical function and quality of life. However, patients have difficulty taking deep breaths due to movement restriction and pain in the postoperative period. Therefore, deep breathing exercises need to be performed regularly to support the incision site in order to ensure effective inspiration and expiration in these patients.

Oxygenation of the traumatized tissues must be sufficient for wound healing in the postoperative incisional area. This oxygen requirement is met by effective ventilation. However, after surgery, patients have difficulty in breathing deeply due to reasons such as pain and limitation of movement. Studies have shown that the practice of planned breathing exercises reduces stress in patients in the pre- and post-operative period, provides calming, and positively affects the level of pain and wound healing. In this respect, planned patient education and care to be given to patients before surgery is very effective in preventing complications related to surgical intervention.

One of the basic duties of surgical nurses is to teach and apply deep breathing and coughing exercises to the patient in pre-operative patient education. It is very important to explain the importance of these exercises to the patient and the effects of performing them at regular intervals on the quality of recovery.

However, studies have drawn attention to the fact that the rates of teaching and applying deep breathing exercises to patients are not at the desired level.

In the literature, many non-pharmacological applications such as acupressure, massage, breathing exercises, listening to music, chewing gum have been performed on patients after surgery and their effects on parameters such as pain, nausea-vomiting, anxiety, vital signs, early discharge, and early mobilization have been examined. There are studies on the relationship between breathing exercises and pain, anxiety, and nausea-vomiting after general surgery surgery, but they are limited. Therefore, the aim of this study is to determine the effect of breathing exercises on pain, anxiety, and nausea-vomiting in patients hospitalized in the general surgery clinic.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and over, Having undergone general surgery with general anaesthesia. They do not have physical/mental disabilities, limitations and diseases that would prevent them from breathing exercises (such as the use of drugs that affect breathing and requiring oxygen therapy, etc.) Cognitive level scales are suitable for application; patients with video phones and no communication problems were included in the study.

Exclusion Criteria:

* Postoperative hemodynamic values unstable, Developing any complications such as severe bleeding, nausea, vomiting after surgery, Leaving work voluntarily, Patients with acute or chronic lung disease were not included in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 149 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
The State-Trait Anxiety Inventory (STAI | 1 day before surgery
  The scale consists of two parts, the 'state anxiety scale', which is created with the aim of determining the instantaneous feelings, and the 20-item 'trait anxiety scale', which was created to determine the feelings in general. It is a four degree scale ranging from 'Nothing' to 'All'. Scores range from 20 (low anxiety) to 80 (high anxiety).
The State Anxiety Inventory (SAI) | On the day of surgery
  The scale consists of two parts, the 'state anxiety scale', which is created with the aim of determining the instantaneous feelings, and the 20-item 'trait anxiety scale', which was created to determine the feelings in general. It is a four degree scale ranging from 'Nothing' to 'All'. Scores range from 20 (low anxiety) to 80 (high anxiety).
The State Anxiety Inventory (SAI) | 1st day after surgery
  The scale consists of two parts, the 'state anxiety scale', which is created with the aim of determining the instantaneous feelings, and the 20-item 'trait anxiety scale', which was created to determine the feelings in general. It is a four degree scale ranging from 'Nothing' to 'All'. Scores range from 20 (low anxiety) to 80 (high anxiety).
The State Anxiety Inventory (SAI) | 15st day after surgery
  The scale consists of two parts, the 'state anxiety scale', which is created with the aim of determining the instantaneous feelings, and the 20-item 'trait anxiety scale', which was created to determine the feelings in general. It is a four degree scale ranging from 'Nothing' to 'All'. Scores range from 20 (low anxiety) to 80 (high anxiety).
The State Anxiety Inventory (SAI) | 30st day after surgery
  The scale consists of two parts, the 'state anxiety scale', which is created with the aim of determining the instantaneous feelings, and the 20-item 'trait anxiety scale', which was created to determine the feelings in general. It is a four degree scale ranging from 'Nothing' to 'All'. Scores range from 20 (low anxiety) to 80 (high anxiety).
Rhodes Nausea and Vomiting Index | 1 day before surgery
  The index's alpha internal consistency coefficient is 0.98, and the alpha internal consistency coefficients for the subgroups range from 0.83 to 0.99. The adaptation of the Rhodes Nausea and Vomiting Index to the Turkish population was done by Genç (2010). In Genç's (2010) adaptation, the internal consistency coefficient was found to be 0.95, with the alpha internal consistency for the subgroups ranging from 0.81 to 0.95. In scoring the "Nausea and Vomiting Index," items 1, 3, 6, and 7 are reverse scored. For each response, 4 indicates the highest level of distress, and 0 indicates the lowest level of distress. The patient's nausea and vomiting experiences for each of the 8 items are summed. The highest possible score is 32, indicating the most severe symptom occurrence.
Rhodes Nausea and Vomiting Index | 1st day after surgery
  The index's alpha internal consistency coefficient is 0.98, and the alpha internal consistency coefficients for the subgroups range from 0.83 to 0.99. The adaptation of the Rhodes Nausea and Vomiting Index to the Turkish population was done by Genç (2010). In Genç's (2010) adaptation, the internal consistency coefficient was found to be 0.95, with the alpha internal consistency for the subgroups ranging from 0.81 to 0.95. In scoring the "Nausea and Vomiting Index," items 1, 3, 6, and 7 are reverse scored. For each response, 4 indicates the highest level of distress, and 0 indicates the lowest level of distress. The patient's nausea and vomiting experiences for each of the 8 items are summed. The highest possible score is 32, indicating the most severe symptom occurrence.
Rhodes Nausea and Vomiting Index | 15st day after surgery
  The index's alpha internal consistency coefficient is 0.98, and the alpha internal consistency coefficients for the subgroups range from 0.83 to 0.99. The adaptation of the Rhodes Nausea and Vomiting Index to the Turkish population was done by Genç (2010). In Genç's (2010) adaptation, the internal consistency coefficient was found to be 0.95, with the alpha internal consistency for the subgroups ranging from 0.81 to 0.95. In scoring the "Nausea and Vomiting Index," items 1, 3, 6, and 7 are reverse scored. For each response, 4 indicates the highest level of distress, and 0 indicates the lowest level of distress. The patient's nausea and vomiting experiences for each of the 8 items are summed. The highest possible score is 32, indicating the most severe symptom occurrence.
Rhodes Nausea and Vomiting Index | 30st day after surgery
  The index's alpha internal consistency coefficient is 0.98, and the alpha internal consistency coefficients for the subgroups range from 0.83 to 0.99. The adaptation of the Rhodes Nausea and Vomiting Index to the Turkish population was done by Genç (2010). In Genç's (2010) adaptation, the internal consistency coefficient was found to be 0.95, with the alpha internal consistency for the subgroups ranging from 0.81 to 0.95. In scoring the "Nausea and Vomiting Index," items 1, 3, 6, and 7 are reverse scored. For each response, 4 indicates the highest level of distress, and 0 indicates the lowest level of distress. The patient's nausea and vomiting experiences for each of the 8 items are summed. The highest possible score is 32, indicating the most severe symptom occurrence.
Brief Pain Inventory | 1 day before surgery
  The Turkish validity and reliability study was conducted by Dicle et al. The Brief Pain Inventory, which has high validity and reliability in different patient groups, has been translated into various languages. This short, simple, and understandable inventory consists of seven items related to the severity of pain and the extent to which pain interferes with daily activities. The pain severity measurements include the worst, least, average, and current pain over the last 24 hours. Pain severity is measured using a numerical pain scale (0 = no pain, 10 = unbearable pain). The dimensions of pain expressed by the individual measure the general activity status, emotional status, relationships with others, walking ability, exercise, sleep, and enjoyment of life due to pain over the past 24 hours. The Cronbach's alpha coefficient was found to be 0.79 for pain severity and 0.80 for the impact of pain.
Brief Pain Inventory | On the day of surgery
  The Turkish validity and reliability study was conducted by Dicle et al. The Brief Pain Inventory, which has high validity and reliability in different patient groups, has been translated into various languages. This short, simple, and understandable inventory consists of seven items related to the severity of pain and the extent to which pain interferes with daily activities. The pain severity measurements include the worst, least, average, and current pain over the last 24 hours. Pain severity is measured using a numerical pain scale (0 = no pain, 10 = unbearable pain). The dimensions of pain expressed by the individual measure the general activity status, emotional status, relationships with others, walking ability, exercise, sleep, and enjoyment of life due to pain over the past 24 hours. The Cronbach's alpha coefficient was found to be 0.79 for pain severity and 0.80 for the impact of pain.
Brief Pain Inventory | 1st day after surgery
  The Turkish validity and reliability study was conducted by Dicle et al. The Brief Pain Inventory, which has high validity and reliability in different patient groups, has been translated into various languages. This short, simple, and understandable inventory consists of seven items related to the severity of pain and the extent to which pain interferes with daily activities. The pain severity measurements include the worst, least, average, and current pain over the last 24 hours. Pain severity is measured using a numerical pain scale (0 = no pain, 10 = unbearable pain). The dimensions of pain expressed by the individual measure the general activity status, emotional status, relationships with others, walking ability, exercise, sleep, and enjoyment of life due to pain over the past 24 hours. The Cronbach's alpha coefficient was found to be 0.79 for pain severity and 0.80 for the impact of pain.
Brief Pain Inventory | 15st day after surgery
  The Turkish validity and reliability study was conducted by Dicle et al. The Brief Pain Inventory, which has high validity and reliability in different patient groups, has been translated into various languages. This short, simple, and understandable inventory consists of seven items related to the severity of pain and the extent to which pain interferes with daily activities. The pain severity measurements include the worst, least, average, and current pain over the last 24 hours. Pain severity is measured using a numerical pain scale (0 = no pain, 10 = unbearable pain). The dimensions of pain expressed by the individual measure the general activity status, emotional status, relationships with others, walking ability, exercise, sleep, and enjoyment of life due to pain over the past 24 hours. The Cronbach's alpha coefficient was found to be 0.79 for pain severity and 0.80 for the impact of pain.
Brief Pain Inventory | 30st day after surgery
  The Turkish validity and reliability study was conducted by Dicle et al. The Brief Pain Inventory, which has high validity and reliability in different patient groups, has been translated into various languages. This short, simple, and understandable inventory consists of seven items related to the severity of pain and the extent to which pain interferes with daily activities. The pain severity measurements include the worst, least, average, and current pain over the last 24 hours. Pain severity is measured using a numerical pain scale (0 = no pain, 10 = unbearable pain). The dimensions of pain expressed by the individual measure the general activity status, emotional status, relationships with others, walking ability, exercise, sleep, and enjoyment of life due to pain over the past 24 hours. The Cronbach's alpha coefficient was found to be 0.79 for pain severity and 0.80 for the impact of pain.

CONTACTS AND LOCATIONS:
Overall Officials: Gamze BULUT ÖZLÜ, Principal Investigator — Ataturk Unıversty
Locations (1):
- Gamze BULUT, Erzurum, Palandöken, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No